CLINICAL TRIAL: NCT03648814
Title: Efficacy and Safety of Intracameral Versus Intravitreal Bevacizumab Injection as an Adjunctive Therapy Before Trabeculectomy With Mitomycin-C in Neovascular Glaucoma: A Prospective Randomized Trial
Brief Title: Intracameral Versus Intravitreal Bevacizumab Injection in NVG: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Assoc. Prof., Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC6100321
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma, Neovascular; Vascular Endothelial Growth Factor Overexpression
Keywords: Neovascular glaucoma
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Intracameral Injection; Intravitreal Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intracameral injection (Experimental): Intracameral Bevacizumab 1.25 mg/0.05 mL. Injection
  Interventions: Procedure: Intracameral injection
- Intravitreal injection (Experimental): Intravitreal Bevacizumab 1.25 mg/0.05 mL. Injection
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intracameral injection — A/C injection of 1.25 mg/0.05 mL bevacizumab
  Arms: Intracameral injection
Procedure: Intravitreal injection — Vitreous injection of 1.25 mg/0.05 mL bevacizumab
  Arms: Intravitreal injection

SUMMARY:
To prospect studying the efficacy and safety of treating NVG with the intracameral versus the intravitreal injection of Bevacizumab.

DETAILED DESCRIPTION:
The present study comparing the safety and efficacy of 1.25mg/0.05mL Bevacizumab injection via the intracameral route versus the intravitreal route in treating the neovascular glaucoma

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of neovascular glaucoma
2. The patients having IOP > 21 mmHg, having the indication for trabeculectomy
3. The patients' age of at least 18-year-old
4. The patients having visual potential at least hand motion.
5. Present of NVI or NVA.
6. Willing and able to provide informed consent to participate in the study
7. Able to understand the purpose of the study, his/her role, and is available to return to the clinic/hospital for all required follow-up visits

Exclusion Criteria:

1. One eye patient
2. Patients having severe corneal edema or total hyphema obscure NVI or NVA view.
3. Cannot obtain endothelial cell count.
4. History of bevacizumab or fluorescence dye allergy.
5. Active infectious ocular disease including endophthalmitis and corneal ulcer
6. History of systemic disease including ischemic heart disease, cerebrovascular disease, end-stage renal disease, liver failure, uncontrolled hypertension
7. Has or planning to be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
regression of nevolascularization | 2 months
  Amount of nevolascular of iris and angle regression

SECONDARY OUTCOMES:
IOP reduction | 2 months
  IOP reduction at 2-month visit compare to baseline
Injection complication | 2 days
  Hyphema, IOP spike

CONTACTS AND LOCATIONS:
Overall Officials: Assoc.Prof.Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Glaucoma unit , Department of Ophthalmology Faculty of Medicine Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No